CLINICAL TRIAL: NCT02105818
Title: Swallowing Difficulties With Medication Intake and Coping Strategies in Patients With Systemic Sclerosis: a Cross-sectional Cohort Study
Brief Title: Swallowing Difficulties With Medication Intake and Coping Strategies in Patients With Systemic Sclerosis
Acronym: SWAMECO
Status: Completed | Type: Observational
Sponsor: Kurt Hersberger (Other)
Collaborators: University of Basel (Other); Reha Rheinfelden (Other)
Responsible Party: Sponsor-Investigator, Kurt Hersberger, Professor, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: SWAMECO_1
Record Dates: First submitted 2014-03-28; First posted 2014-04-07 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Systemic Sclerosis; Deglutition Disorders; Adherence to Medication Regime; Coping Behaviour; Scleroderma, Systemic
Keywords: Self-reported questionnaire; Swallowing disorders; Systemic sclerosis; Drug therapy; Adherence to medication regime; Coping strategy; Pharmaceutical care; Patient safety; Patient oriented care
MeSH Terms: conditions — Scleroderma, Systemic; Deglutition Disorders; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Systemic sclerosis: Patients with diagnosed systemic sclerosis treated in the Reha Rheinfelden, Switzerland (European Centre for the Rehabilitation of Scleroderma).

SUMMARY:
The purpose of this study is the validation of a newly developed self-report questionnaire which aims at determining the prevalence, location and intensity of SWAllowing difficulties with drug intake, and describing the impact on MEdication regimen focusing on COping strategies (SWAMECO).

DETAILED DESCRIPTION:
The study aims at investigating a cohort of patients with diagnosed systemic sclerosis using the newly developed self-report SWAMECO-questionnaire.

The self-report questionnaire is sub-divided into four sections: detection of swallowing difficulties, coping strategies, risk factors to develop swallowing difficulties and adherence to medication.

This study involves patients with systemic sclerosis. Systemic sclerosis often is accompanied by swallowing disorders which may lead to issues in handling medication regimen with risks for patient safety.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* diagnosis for systemic sclerosis
* treated in the Reha Rheinfelden
* signed informed consent
* german language skills

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed systemic sclerosis treated in the Reha Rheinfelden, Switzerland (European Centre for the Rehabilitation of Scleroderma)
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Validation of the SWAMECO self-report questionnaire | Eligible patients will be asked to answer the questionnaire at the time of enrolment (cross-sectional), return of all questionnaires within 4 weeks.
  Face validation of the questionnaire in a convenience sample of patients with systemic sclerosis.
  Percentage of patients who are able to fill out the SWAMECO questionnaire completely and correctly regarding the different types of scales (visual-analog-scale, likert-scale), dichotomous questions (yes / no), and figures to describe symptoms.

SECONDARY OUTCOMES:
Location and intensity of swallowing difficulties | Eligible patients will be asked to answer the questionnaire at the time of enrolment (cross-sectional), return of all questionnaires within 4 weeks.
  Patients describe location and intensity of swallowing difficulties with medication intake by filling the SWAMECO self-report questionnaire
Coping strategies | Eligible patients will be asked to answer the questionnaire at the time of enrolment (cross-sectional), return of all questionnaires within 4 weeks.
  Patients describe coping strategies to avoid swallowing difficulties with medication intake by filling the SWAMECO self-report questionnaire
Adherence to medication regimen | Eligible patients will be asked to answer the questionnaire at the time of enrolment (cross-sectional), return of all questionnaires within 4 weeks.
  Patients describe adherence to medication regimen using the Morisky 8-Item Medication Adherence Questionnaire (MMAS-8).
Prevalence of present and/or past swallowing difficulties with medication intake | Eligible patients will be asked to answer the questionnaire at the time of enrolment (cross-sectional), return of all questionnaires within 4 weeks.
  Patients describe present and/or past swallowing difficulties with medication intake by filling the SWAMECO self-report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Hersberger, Prof, Study Chair — Pharmaceutical Care Research Group, University of Basel, Switzerland; Markus Messerli, MSc, Study Director — Pharmaceutical Care Research Group, University of Basel, Switzerland; Michael Buslau, PD MD, Principal Investigator — Reha Rheinfelden, Switzerland; Rebecca Wysser, BSc, Principal Investigator — Pharmaceutical Care Research Group, University of Basel, Switzerland; Isabelle Arnet, PhD, Principal Investigator — Pharmaceutical Care Research Group, University of Basel, Switzerland
Locations (1):
- Reha Rheinfelden, Rheinfelden, Canton of Aargau, Switzerland

REFERENCES:
- [Background] Marquis J, Schneider MP, Payot V, Cordonier AC, Bugnon O, Hersberger KE, Arnet I. Swallowing difficulties with oral drugs among polypharmacy patients attending community pharmacies. Int J Clin Pharm. 2013 Dec;35(6):1130-6. doi: 10.1007/s11096-013-9836-2. Epub 2013 Aug 21. PMID 23963541
- [Background] Schiele JT, Quinzler R, Klimm HD, Pruszydlo MG, Haefeli WE. Difficulties swallowing solid oral dosage forms in a general practice population: prevalence, causes, and relationship to dosage forms. Eur J Clin Pharmacol. 2013 Apr;69(4):937-48. doi: 10.1007/s00228-012-1417-0. Epub 2012 Sep 29. PMID 23052416
- See also: Homepage of the Pharmaceutical Care Research Group, University of Basel, Switzerland — http://www.pharmacare.unibas.ch